CLINICAL TRIAL: NCT07080684
Title: Short-Term Dual Antiplatelet Therapy With Early Transition to Low-dose Antiplatelet Monotherapy Using ticagRelor in Chronic Coronary Artery Disease
Brief Title: Short-Term Dual Antiplatelet Therapy With Early Transi-tion to Low-dose Antiplatelet Monotherapy Using Ti-cagRelor in Chronic Coronary Artery Disease
Acronym: STELAR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Rodolfo Caminiti, Principal Investigator, Interventional Cardiologist, University of Messina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STELAR_CCS_0725
Record Dates: First submitted 2025-07-03; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Chronic Coronary Syndrome
MeSH Terms: interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short DAPT with Ticagrelor 60 mg (Experimental): * 1-month DAPT: aspirin + ticagrelor 60 mg BID
  * Followed by 5-month ticagrelor 60 mg BID monotherapy
  * Ticagrelor will be provided by the sponsor (off-label use)
  Interventions: Drug: Ticagrelor 60 mg
- Standard DAPT with Clopidogrel (Active Comparator): - 6-month DAPT: aspirin + clopidogrel 75 mg daily
  Interventions: Drug: clopidogrel 75 mg

INTERVENTIONS:
Drug: Ticagrelor 60 mg — Patients in this arm will receive dual antiplatelet therapy (DAPT) consisting of low-dose ticagrelor (60 mg twice daily) plus aspirin (75-100 mg once daily) for 1 month, followed by ticagrelor 60 mg monotherapy for 5 additional months (total 6 months of therapy).
  This strategy aims to reduce ischemic events while minimizing bleeding risk by leveraging the potent antiplatelet effect of ticagrelor at a lower maintenance dose.
  Arms: Short DAPT with Ticagrelor 60 mg
Drug: clopidogrel 75 mg — Patients in the control group will receive standard DAPT consisting of clopidogrel 75 mg once daily plus aspirin 75-100 mg once daily for 6 months.
  This represents the current standard of care in patients with chronic coronary syndrome (CCS) undergoing percutaneous coronary intervention (PCI) with drug-eluting stents.
  Arms: Standard DAPT with Clopidogrel

SUMMARY:
This is a prospective, multicenter, randomized, open-label trial with blinded endpoint adjudication (PROBE design), comparing one-month dual antiplatelet therapy (DAPT) with low-dose ticagrelor (60 mg BID) followed by ticagrelor monotherapy to standard 6-month DAPT with aspirin and clopidogrel in patients with chronic coronary syndrome (CCS) undergoing percutaneous coronary intervention (PCI). The primary endpoint is a composite of cardiovascular death, all-cause death, myocardial infarction, disabling stroke, target lesion revascularization (TLR), and major bleeding. The study aims to evaluate whether the short DAPT strategy reduces ischemic events while maintaining bleeding safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of informed consent.
* Diagnosis of chronic coronary syndrome (CCS) according to ESC guidelines.
* Undergoing successful PCI with implantation of one or more new-generation drug-eluting stents (DES).
* Indication for dual antiplatelet therapy (DAPT) following PCI.
* Willingness and ability to comply with all study procedures and follow-up assessments.
* Signed informed consent prior to any study-specific procedure.
* Creatinine clearance ≥30 mL/min, calculated using the Cockcroft-Gault formula.
* Life expectancy greater than 1 year in the investigator's judg-ment.
* Hemodynamically stable at the time of randomization.
* Acceptable bleeding risk profile: patients fulfilling ARC-HBR criteria may be included only if the treating physician deems a 6-month antiplatelet regimen to be safe.
* No contraindications to study drugs, including aspirin, clopi-dogrel, or ticagrelor.

Exclusion Criteria:

* Presentation with acute coronary syndrome (ACS), including STEMI, NSTEMI, or unstable angina within the previous 6 mon-ths.
* Planned staged PCI or revascularization procedure within 6 months after index PCI.
* Requirement for long-term oral anticoagulation therapy, such as for atrial fibrillation, mechanical heart valves, or venous thromboembolism.
* History of major bleeding, including gastrointestinal or intra-cranial bleeding, within the past 6 months.
* Severe hepatic impairment, active liver disease, or transamina-ses >3× upper limit of normal.
* Known platelet disorder, coagulopathy, or thrombocytopenia (<100,000/mm³).
* Contraindication or hypersensitivity to aspirin, clopidogrel, or ticagrelor, or known drug interaction that precludes their use.
* Ongoing active bleeding or high risk of bleeding that, in the opinion of the investigator, precludes DAPT.
* Pregnancy or breastfeeding, or women of childbearing potential who are not using effective contraception.
* Life expectancy <1 year due to non-cardiovascular comorbidi-ties (e.g., cancer, advanced renal failure).
* Participation in another interventional clinical trial that may interfere with the outcomes of this study.
* Severe anemia (hemoglobin <9 g/dL) not corrected before ran-domization.
* Inability or unwillingness to provide informed consent or ad-here to study follow-up.
* Prior stroke with residual neurological deficit or history of di-sabling stroke (mRS ≥3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiovascular death, myocardial infarction, disabling stroke, target lesion revascularization, major bleeding, and all-cause death | 6 month
  Number of participants experiencing any of the following events within 12 months after the index percutaneous coronary intervention (PCI):
  * Cardiovascular death - Number of participants with death due to a cardiovascular cause
  * Non-fatal myocardial infarction - Number of participants with myocardial infarction as defined by the Fourth Universal Definition
  * Non-fatal disabling stroke - Number of participants with stroke resulting in a modified Rankin Scale (mRS) ≥2
  * Target lesion revascularization (TLR) - Number of participants undergoing clinically driven revascularization of the target lesion
  * Major bleeding - Number of participants experiencing major bleeding events defined as BARC type 3 or 5
  * All-cause death - Number of participants who died from any cause

SECONDARY OUTCOMES:
Cardiovascular Death | 6 month
  death due to myocardial infarction, sudden cardiac death, stroke, heart failure, or other vascular causes, as adjudicated by investigators.
All cause death | 6 month
  death from any cause, cardiovascular or non-cardiovascular.
Myocardial Infarction | 6 month
  Defined according to ARC-2 criteria as either spontaneous (type 1), peri-procedural (type 4a/4b), or stent thrombosis-related, confirmed by clinical symp-toms, ECG changes, and biomarker elevation.
Major Bleeding (BARC ≥3) | 6 month
  Bleeding events classified as Bleeding Academic Research Consortium (BARC) type 3a (overt bleeding with hemoglobin drop ≥3 g/dL), 3b (requiring in-tervention or surgery), 3c (intracranial or intraocular), or type 5 (fatal bleeding).
Disabling Stroke | 6 month
  New-onset neurologic deficit confirmed by imaging and persisting beyond 24 hours, with a modified Rankin Score (mRS) ≥2.
Target Lesion Revascularization (TLR) | 6 month
  Repeat revascularization (PCI or CABG) of the originally treated lesion due to restenosis or thrombosis.
Target Vessel Revascularization (TVR) | 6 month
  Any repeat PCI or CABG of the same vessel previously treated, regardless of lesion location.
Any Ischemic Event | 6 month
  Composite of MI, ischemic stroke, or TLR.